CLINICAL TRIAL: NCT01184040
Title: Extending Contingency Management's Benefits With Progressively Increasing Variable Interval Prize Reinforcement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-249-1; 1P30DA023918-01A1 (NIH)
Record Dates: First submitted 2010-08-10; First posted 2010-08-18 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Exercise; Addictive Behaviors
MeSH Terms: conditions — Motor Activity; Behavior, Addictive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- (A) Non-contingent control (No Intervention): Participants assigned to the control condition will be told to wear the pedometer daily and select a twice-weekly meeting schedule with research staff for 12 weeks (study weeks 4-15). On days randomly selected as meeting days, participants will be asked to bring in their pedometers. Participants who attend their scheduled meetings will receive a $5 gift card just for attending and bringing the pedometer, so long as it has registered steps walked in at least the past 4 days. They will be congratulated if they walked 10,000 steps or more on the prior 4 days, and encouraged to walk 10,000 steps or more per day on subsequent days.
- VIP CM (Experimental): Participants assigned to Increasing Variable Interval Prize (VIP) Reinforcement group will be scheduled for the same study visits as those in the Control group, but will also earn chances to win prizes if they have walked more than 10,000 steps in the past 4 days.
  Interventions: Behavioral: VIP CM

INTERVENTIONS:
Behavioral: VIP CM — Participants will receive progressively increasing CM for walking 10,000 steps per day over 4 days prior to visit as verified by the pedometer.
  Arms: VIP CM

SUMMARY:
Contingency Management (CM) is highly effective in promoting recovery from substance use disorders, but benefits tend to attenuate over time when CM is discontinued. Identifying modifications of CM delivery that can extend its benefits is an important goal. The goal of this study is to evaluate the use of reinforcements to increase physical activity, specifically walking. The study provides a standard CM intervention to promote walking for three weeks. After three weeks, a progressively increasing variable interval schedule of reinforcement will be evaluated for increasing the durability of effects of the initial CM intervention. We hypothesize that Variable Interval Prize Contingency Management will result in greater adherence to a walking goal of 10,000 steps per day at Week 15 and Week 24 compared to the Control Condition.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* currently not physically active
* Physically able and willing to walk 10,000 steps per day

Exclusion Criteria:

* psychiatric or physical illness that could interfere with participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-05; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
number of steps walked in seven days prior to follow up assessment, as verified by the pedometer | week 15
number of steps walked in seven days prior to follow up assessment, as verified by the pedometer | week 24

CONTACTS AND LOCATIONS:
Overall Officials: Nancy M Petry, Ph.D., Principal Investigator — UConn Health
Locations (1):
- UConn Heatlh Center, Farmington, Connecticut, United States